CLINICAL TRIAL: NCT07088614
Title: Effectiveness of Remote Respiratory Physiotherapy Using a Digital Platform on the Frequency of Exacerbations, Lung Function and Quality of Life, Assessed Before and After 6 Months of Intervention, in Children Aged 6-18 Years With Cystic Fibrosis at Dr. Luis Calvo Mackenna Hospital: a Pre-experimental Study.
Brief Title: Effectiveness of Respiratory Physiotherapy on Frequency of Exacerbations, Lung Function and Quality of Life After 6 Months in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Collaborators: Luis Calvo Mackenna Children´s Hospital (Other)
Responsible Party: Principal Investigator, Andrea Mendez, Full Professor, School of Physiotherapy, Faculty of Health and Social Sciences, University of Americas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DI20/22
Record Dates: First submitted 2025-07-11; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Physiotherapy; Telehealth; Telemedicine; Children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Pre-experimental design, single-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote physiotherapy group (Experimental): Remote respiratory physiotherapy protocol supervised 3 times a week via digital video conference, based on Chilean national guidelines for cystic fibrosis.
  Each 1-hour session (3×/week for 6 months) includes:
  Evaluation: respiratory assessment, teaching and reinforcement of airway clearance techniques, inhaled medication use, physical activity, and adherence to non-physiotherapy care. Six checklists are used to guide and monitor weekly patient activities.
  Respiratory physiotherapy: conducted on-screen by the patient or caregiver, guided remotely. Includes: short-acting bronchodilator (if indicated), 7% hypertonic saline nebulization (10 min), 5-min Flutter/Acapella, ELTGOL or ELPr (2×5 min), and assisted coughing.
  Re-evaluation: reassessment with the initial checklist, Q&A, and scheduling the next session.
  Participants continue their usual hospital-based care and receive baseline and post-intervention measurements.
  Interventions: Other: Remote respiratory physiotherapy

INTERVENTIONS:
Other: Remote respiratory physiotherapy — Remote respiratory physiotherapy protocol supervised 3 times a week via digital video conferencing, based on Chilean national guidelines for cystic fibrosis.
  Each 1-hour session (3×/week for 6 months) includes:
  Evaluation: respiratory assessment, teaching and reinforcement of airway clearance techniques, inhaled medication use, physical activity, and adherence to non-physiotherapy care. Six checklists are used to guide and monitor weekly patient activities.
  Respiratory physiotherapy: conducted on-screen by the patient or caregiver, guided remotely. Includes: short-acting bronchodilator (if indicated), 7% hypertonic saline nebulization (10 min), 5-min Flutter/Acapella, ELTGOL or ELPr (2×5 min), and assisted coughing.
  Re-evaluation: reassessment with the initial checklist, Q&A, and scheduling the next session.
  Participants continue their usual hospital-based care and receive baseline and post-intervention measurements.

SUMMARY:
Daily respiratory physiotherapy is a fundamental part of cystic fibrosis treatment, however, patients adherence is low. Thus, there is a need for studies that evaluate the impact of physiotherapy supervision in patients with cystic fibrosis (CF), with particular emphasis on the effectiveness of telemonitoring. A quantitative, pre-experimental, single-centre study was designed involving the universe of patients with CF from Dr. Luis Calvo Mackenna Hospital to measure frequency of exacerbations, pulmonary function and quality of life, before and after remote respiratory physiotherapy intervention via videoconference platform for 6 months.

DETAILED DESCRIPTION:
This study evaluated the effectiveness of remote respiratory physiotherapy delivered via a videoconferencing platform for children aged 6 to 18 years with cystic fibrosis, who were followed at Dr. Luis Calvo Mackenna Hospital. Cystic fibrosis is a chronic respiratory disease that requires interdisciplinary management from the time of diagnosis, with respiratory physiotherapy being a cornerstone of treatment. Despite its importance, adherence is often low, especially for home-based care. Therefore, the study aimed to determine whether remote supervision could improve key clinical outcomes such as exacerbation frequency, pulmonary function, and quality of life.

The study followed a quantitative, pre-experimental, single-center design, with a non-probabilistic convenience sample. Although the initial target sample size was 16, the final study population included 9 patients, all diagnosed through a sweat test and enrolled in the National Cystic Fibrosis Program. The intervention consisted of remote respiratory physiotherapy sessions, held three times per week for six months, led by a physiotherapist via videoconference. Each session included clinical assessment, airway clearance techniques, supervised use of inhaled medications, physical exercise, and general health education.

Outcomes were measured before and after the intervention. Primary outcomes included the frequency of respiratory exacerbations. Secondary outcomes were lung function (measured by FEV1 and FVC), health-related quality of life (assessed using the PedsQL™ questionnaire), exercise capacity (via the six-minute walk test), days of hospitalization and antibiotic use, treatment adherence, and adverse events. All measurements were performed by trained, blinded professionals according to established clinical standards.

Statistical analysis was conducted using STATA version 14.2. Data distribution was assessed to select appropriate tests: paired t-tests or Wilcoxon tests were used for continuous variables, and McNemar's test was applied to categorical variables. A significance level of 0.05 was used, and results were presented with 95% confidence intervals. All adverse events were documented, including their characteristics, resolution, severity, and potential relation to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cystic fibrosis aged 6 to 18 years.
* Patients admitted to the National Cystic Fibrosis Programme.
* Patients followed at the pulmonology outpatient clinic of Dr. Luis Calvo Mackenna Hospital.

Exclusion Criteria:

* Patients currently undergoing pulmonary rehabilitation.
* Patients undergoing lung transplantation.
* Patients with severe comorbidity affecting survival.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Exacerbations frequency | Frequency of respiratory exacerbations will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  Frequency of respiratory exacerbations over six months expressed as proportion of subjects with <1 exacerbation, 1-2 exacerbations, or >2 exacerbations), using the medical record.

SECONDARY OUTCOMES:
Health-related quality of life | Health-related quality of life will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  Quality of life will be assessed using the PedsQL™ Generic Core Scales, a 23-item generic health-related quality of life questionnaire designed for healthy children and adolescents aged 2-18 years, as well as those with chronic health conditions. The PedsQL™ Young Child Report (ages 5-7), Child Report (8-12), Teen Report (13-18), and corresponding parent proxy reports will be used. The PedsQL™ evaluates four domains: physical, emotional, social, and school functioning, using a 5-point Likert scale, with scores ranging from 0 to 92, where lower scores indicate better health-related quality of life. The PedsQL™ is a valid and reliable instrument, with an internal consistency coefficient of 0.88, and has been used in studies of patients with cystic fibrosis.
FEV1 | FEV1 will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  FEV1 as a percentage of predicted assessed by spirometry using a laboratory spirometer at Dr. Luis Calvo Mackenna Hospital, previously calibrated, following the American Thoracic Society/European Respiratory Society (ATS/ERS) clinical guidelines.
Days of hospitalization | Days of hospitalization will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  Days of hospitalization will be assessed using the medical record as number of days
Days on intravenous/oral antibiotic treatment for respiratory causes | Days on intravenous/oral antibiotic treatment will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  Days on intravenous/oral antibiotic treatment for respiratory causes will be assessed in the last 6 months, using the medical record.
Exercise capacity | Exercise capacity will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  Exercise capacity will be assessed using the 6-Minute Walk Test (6MWT), a reliable and valid test to measure exercise tolerance in children with cystic fibrosis. During the test, oxygen saturation (SpO₂) and heart rate (HR) will be continuously monitored and recorded at the beginning and end of the test, using the patient's own pulse oximeter or one provided by the study. Dyspnea will be assessed using the modified Borg scale at the beginning and end of the test. The exercise capacity will be expressed as distance walked, in meters,
Treatment adherence | Treatment adherence will be assessed at the end of the study, i.e. six months after the beginning of the intervention.
  Treatment adherence will be determined as the percentage of compliance with the intervention guidelines.
Adverse events | The occurrence of adverse events will be assessed from the beginning of the intervention up to six months after the beginning of the intervention.
  The occurrence of adverse events will be assessed using the medical record.
FVC | FVC will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  FVC as a percentage of predicted by spirometry using a laboratory spirometer at Dr. Luis Calvo Mackenna Hospital, previously calibrated, following the American Thoracic Society/European Respiratory Society (ATS/ERS) clinical guidelines.
FEV1/FVC | FEV1/FVC will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention, and at the end of the study, i.e. six months after the beginning of the intervention.
  FEV1/FVC as a percentage assessed by spirometry using a laboratory spirometer at Dr. Luis Calvo Mackenna Hospital, previously calibrated, following the American Thoracic Society/European Respiratory Society (ATS/ERS) clinical guidelines.

OTHER OUTCOMES:
Age | Age will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Age expressed in years will be determined using the medical record
Sex | Sex will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Sex will be expressed as female or male, and it will be determined using the medical record
Age at diagnosis | Age at diagnosis will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Age at diagnosis expressed in years will be determined using the medical record
Body Mass Index (BMI) | Body Mass Index (BMI) will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Body Mass Index (BMI) will be calculated using the weight-to-height ratio (weight in kilograms/height in meters), both measured by stadiometer and scale.
Co-morbidity | Co-morbidity will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Co-morbidity will be determined using the medical record
Frequency of outpatient physiotherapy visits | Frequency of outpatient physiotherapy visits will be assessed at the baseline, 2 weeks maximum before the beginning of the intervention
  Frequency of outpatient physiotherapy visits will be expressed as times/month, and it will be determined using the medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Luis Calvo Mackenna Children's Hospital, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Because it has not been required by other researchers.

REFERENCES:
- [Background] Lavie M, Vilozni D, Sokol G, Somech R, Szeinberg A, Efrati O. Hospital versus home treatment of respiratory exacerbations in cystic fibrosis. Med Sci Monit. 2011 Dec;17(12):CR698-703. doi: 10.12659/msm.882129. PMID 22129901
- [Background] Goodfellow NA, Hawwa AF, Reid AJ, Horne R, Shields MD, McElnay JC. Adherence to treatment in children and adolescents with cystic fibrosis: a cross-sectional, multi-method study investigating the influence of beliefs about treatment and parental depressive symptoms. BMC Pulm Med. 2015 Apr 26;15:43. doi: 10.1186/s12890-015-0038-7. PMID 25927329
- [Background] Thornton J, Elliott R, Tully MP, Dodd M, Webb AK. Long term clinical outcome of home and hospital intravenous antibiotic treatment in adults with cystic fibrosis. Thorax. 2004 Mar;59(3):242-6. doi: 10.1136/thx.2003.005876. PMID 14985563